CLINICAL TRIAL: NCT04692623
Title: EFFECTS OF MOXIFLOXACIN AND GEMIFLOXACIN ON BLOOD GLUCOSE LEVEL OF EUGLYCEMICS:A PRE-CLINICAL AND CLINICAL STUDY
Brief Title: EFFECTS OF MOXIFLOXACIN AND GEMIFLOXACIN ON BLOOD GLUCOSE AND ECG MORPHOLOGY OF EUGLYCEMICS:A CLINICAL STUDY
Acronym: CT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaheed Benazir Bhutto University Sheringal Dir Upper (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Dr Shujaat Ahmad, Associate Professor in Pharmacy,SBBU,Sheringal Dir Upper, Shaheed Benazir Bhutto University Sheringal Dir Upper
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: ShaheedBBUSheringalD
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Blood Glucose, Low; Hypoglycemia
Keywords: ,Blood glucose,Serum insulin
MeSH Terms: conditions — Hypoglycemia | interventions — Moxifloxacin; Blood Glucose; Gemifloxacin

STUDY DESIGN:
Intervention Model Description: Single group for Moxifloxacin having 30 healthy euglycemic volunteers, another group for Gemifloxacin having 30 healthy euglycemic volunteers
Who Masked: Participant, Investigator
Masking Description: Proper care shall be taken while taking blood samples for checking blood glucose and serum insulin levels as per ICH good clinical practices guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moxfloxacin Group (Experimental): In this arm 30 healthy volunteers were selected and they were given Moxifloxacin drug.
  Interventions: Drug: Moxifloxacin 400mg
- Gemifloxacin Group (Experimental): In this arm 30 healthy volunteers were selected and they were given Gemifloxacin
  Interventions: Drug: Gemifloxacin 320 MG

INTERVENTIONS:
Drug: Moxifloxacin 400mg — Blood will be checked for glucose levels and ECG at Baseline(Day Ist) and at Steady state Steady state(Tmax) via Glucometer and ECG machine will be used for determination of serum insulin levels.
  Other Names: Blood glucose and serum insulin
  Arms: Moxfloxacin Group
Drug: Gemifloxacin 320 MG — Blood will be checked for glucose levels and ECG at Baseline(Day Ist) and at Steady state(Tmax) via Glucometer and ECG machine will be used for determination of serum insulin levels.
  Other Names: Blood glucose and serum insulin
  Arms: Gemifloxacin Group

SUMMARY:
EFFECTS OF MOXIFLOXACIN AND GEMIFLOXACIN ON BLOOD GLUCOSE LEVEL OF EUGLYCEMICS:A PRE-CLINICAL AND CLINICAL STUDY.

Our aim and objectives are to:

1. To check the possible effects of Moxifloxacin and Gemifloxacin in healthy volunteers for possible effects on blood glucose levels with a subsequent shift in serum insulin level of healthy volunteer (target population).
2. ECG morphology effect. In the above entitled studies we are going to determine the effects of the above two 4th generation fluoroquinolones drugs on the blood glucose levels and ECG morphology effect.of euglycemics healthy volunteers.The drug will be gave as per approved standard adult dose.The drug is FDA approved and marketed drug.No risk is to the patient only 3-5 ml of the blood will be taken at baseline and after the drug completion at steady state concentration.

DETAILED DESCRIPTION:
The study will be conducted under good clinical practice guidelines and a consent form will be signed from the healthy volunteers as per design of World health organization.The study has no harmful effects on the heaths of the volunteers as we are conducting the study for five dose/one pack drug will be gaven. The volunteers will be sampled randomly and the effect of the said drugs will be determined on blood glucose and insulin level.

Diabetes mellitus (DM), a non-communicable disease, which is considered now-a-days a life threatening disease to the human health (1,2).According to the report of International Diabetes Federation (IFD) and World Health Organization (WHO), diabetes mellitus is one of the World's fifth leading cause of mortality and about 415 million people of the world's population have diabetes mellitus in 2018 (3). After every 6 seconds, a person dies from diabetes mellitus (4, 5). Pakistan is a country with 7th highest diabetic population in the world and it is assumed to rise to 4th highest place by 2030 (6). Due to sedentary life style of People, there is a maximum increase of DM in the last decade (7). DM is classified into two classes i.e. Type I and Type II (8). The Type I diabetes is much more common. It is due to defective insulin secretion or insulin action or both (9). The Type II diabetes is now-a-days attributed to genetic disorders affecting the beta cells of the pancreas (10), or the ability of body cells to respond to insulin action leading to insulin resistance DM (11, 12).

Fluoroquinolones (FQs) are a group of antibacterial antibiotics. Newer fluoroquinolones has expanded its traditional coverage from Gram-negative coverage to Gram-positive as well as to anaerobic organisms (14-16). It has been used since 2-3 decades and has been observed to have excellent anti-microbial coverage, but unfortunately the FQs are associated with adverse drug events including strong dysglycemic effects which has also led to irreversible brain damage and even death (17). Till date, six different types of adverse drug reactions have been reported with Fluoroquinolones. These include prolongation of QT interval, Photo toxicity, hepatotoxicity and alteration in the blood glucose hemostasis (hyperglycemia or sometimes hypoglycemia), damage to the tendons leading to tendinitis (18). Canadian Adverse Drug Reaction Monitoring Program (CADRMP) reported that three marketed fluoroquinolones namely gatifloxacin, levofloxacin and moxifloxacilin are under Metabolic and Nutritional Disorders category. Among them Temafloxacin, levofloxacin and gatifloxacin have been reported to be associated with hemolysis (19).

It has been assumed that the dysglycemic effects of FQs mainly occur through their action on the ATP- sensitive K + channels. According to definition, an agent that causes the selective relaxation of an induced contractility due to low K+ (20-25 mM) is grouped as K+ channel opener. From the studies it can be assumed that fluoroquinolones may block the ATP-sensitive K+ channels as well as the opening of as Calcium channels that are voltage dependent (22). These opened Calcium channels further depolarize the membrane potential ultimately releasing insulin. These Studies reveals that fluoroquinolones have pancreatic beta cell cytotropic activity, however the dysglycemic effects of Moxifloxacin and Gemifloxacin have not been proven but very strong associations have been demonstrated via some case report studies (21).

Keeping in view all these studies and developments regarding the adverse effects associated with fluoroquinolones specially the dysglycemic effects due to cytotropic influence on the beta cells of the pancreas it is now very much needed to actually correlate these effects seen in the beta cells of the pancreas with the pancreatic tissue histopathological changes. Since, Moxifloxacin and Gemifloxacin are a new generation quinolones, thus our study focuses on them to get a clear picture of its possible shift of blood glucose and insulin in our society. Thus the hallmark of our study is to focus on dysglycemic effects (either hyperglycemic or hypoglycemic effects) associated with quinolones, it is not clear to get a clear picture on blood glucose level until it is tested in control environment of a preclinical study, and to translate the possible effects of the preclinical study in a controlled clinical trial of healthy volunteers who are euglycemics as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers having age from 20- 40 years
* Non-Diabetic
* Non-Alcoholics
* Non-Smokers
* Non-Hypertensive

Exclusion Criteria:

* Patients with QT interval prolongation in ECG
* Patients unwilling to give consent
* Patients already on antibiotic therapy for a period one to two week or above.
* Patients who are on other drugs that induces or decreases drug metabolism of quinolones.
* Pregnant female patients.
* Abuse of alcoholic beverages
* Participants who are Allergic or Hypersensitivity to the said drug
* Participants who have participated in a clinical trial within 3 months before the study period.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both male and female healthy euglycemic volunteers are eligible for inclusion in the studies
Enrollment: 25 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia expected as per case reports and studies | 4 weeks
  Blood glucose level monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Abid Ullah, Ph.D Scholar, Study Chair — Departemt of Pharmacy,Shaheed Benazir Bhutto University,Sheringal Dir Upper,KP,Pakistan
Locations (1):
- Khyber Medical University,Peshawar, Peshawar, Khyber Pukhtan Khawa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The data once obtained will be published in reputed journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one month for complete data cllection and compilation
Access Criteria: At the official website of Shaheed Benazir Bhutto University sheringal Dir upper
URL: http://www.sbbu.edu.pk

REFERENCES:
- [Background] Zimmet P. Globalization, coca-colonization and the chronic disease epidemic: can the Doomsday scenario be averted? J Intern Med. 2000 Mar;247(3):301-10. doi: 10.1046/j.1365-2796.2000.00625.x. PMID 10762445
- [Derived] Ullah A, Ahmad S, Ali N, Rahman SU, Hussain H, Alghamdi S, Almehmadi M, Dablool AS, Bannunah AM, Bukhari SH, Almarshad F. Insulinotropic Potential of Moxifloxacin and Gemifloxacin: An In Vivo Rabbits Model Study Followed by Randomized Phase I Clinical Trial. Antibiotics (Basel). 2022 Jan 24;11(2):148. doi: 10.3390/antibiotics11020148. PMID 35203750